CLINICAL TRIAL: NCT02042326
Title: Prospective Evaluation of the Efficacy of Sirolimus (Rapamune®) in the Treatment of Severe Arteriovenous Malformations
Acronym: MAV-RAPA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRCN10-PR-DEVAUCHELLE; 2011-000321-69 (EudraCT Number)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Arteriovenous Malformations
Keywords: Arteriovenous Malformations; Sirolimus; Maxillofacial Surgery
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus treatment (Experimental): Patients will receive sirolimus (Rapamune). The dose should be adjusted to obtain a residual plasma rate of 8 to 12 ng/ml in 4 weeks. This serum level will be maintained throughout the duration of the study in the absence of side effects. In case of intolerance that do not justify the discontinuation of treatment, the dose may be reduced by maintaining a serum level greater than 3 ng/ml.
  The starting dose will be 2 mg per day, and will be adapted every week for one month.
  The preferred dosage form is tablet form. To prevent common side effects in early treatment, corticosteroids based prednisolone (SOLUPRED) will be established at a dose of 0.5 mg/ kg/day for the first week of treatment.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — For patients with swallowing problems, and for children under 6 years and / or who have an inability to swallow tablets, the 1mg/ml solution form should be used.
  Other Names: Rapamune

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of sirolimus (oral form), to decrease the volume and symptoms due to superficial arteriovenous malformations (AVM).

Sirolimus has properties that reduce the activity of the immune system (immunosuppressant), to fight against the proliferation of cancer cells (anti- tumor) and also reduce the proliferation of blood vessels (anti -vascular). Sirolimus is primarily used in transplant patients to prevent organ transplant rejection. Many animal and laboratory studies were carried out and demonstrate in particular the activity of sirolimus on vessels. It is this anti- vascular effect that could help treat arteriovenous malformations.

DETAILED DESCRIPTION:
Anti-proliferative and anti-angiogenic properties of Sirolimus (Rapamycin®) are the basis of the rationale to use it in the treatment of arteriovenous malformations, for which the pathophysiology remains poorly understood. The interest of this class of drug is that inhibition of mTOR (mammalian target of rapamycin) may also block growth and / or angiogenic factors (other than VEGF) involved in the development of AVM. More specifically anti-VEGF drugs does not have that potential.

ELIGIBILITY:
Inclusion Criteria:

* Patients (adults, adolescents and children older than 2 years), with arteriovenous malformation stage II + III or IV (according to Schöbinger's classification) : active or quiescent, marked or not by hemorrhagic phenomena.
* Patients (parents for minors) must sign a consent form established after clear information risks and expected benefits of the study.
* Patients (major and minor of childbearing age) must have effective contraception during the study period and continuing until 12 weeks after the end of treatment
* Negative pregnancy blood test for women of childbearing age.

Exclusion Criteria:

* Chronic or acquired immunosuppression :

  * patients with transplanted organ or who received a hematopoietic stem cell
  * patient with congenital immunodeficiency
* Patients implanted with chronic active infection associated with hepatitis B , hepatitis C or HIV
* Pregnant or nursing woman.
* Allergy to macrolides
* Allergy to peanut or soya
* Hypersensitivity to " Sirolimus " or any of the excipients of the investigational product
* Contraindications to performing an MRI
* Leukopenia below 1 000 /mm3
* Thrombocytopenia lower to 80,000 /mm3
* Anemia with Hb < 9 g/dl
* Elevated transaminase > 2.5 N
* History of cancer less than two years before the inclusion
* Surgery older than 2 months before inclusion
* Active infection (viral and bacterial ) on the date of inclusion
* Hypercholesterolemia > 7 mmol / l despite appropriate medical treatment
* Hyperlipidemia > 2 mmol / l despite appropriate medical treatment
* Uncontrolled diabetes
* Patients unable to follow a clinical study
* Major under guardianship, persons deprived of their liberty

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09-12 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy at M12 | After 12 months of treatment
  The efficacy of treatment is a composite criteria based on:
  * The proportion of patients with no evolution of the AVM during the study period,
  * The proportion of patients with a reduction in tumor volume of the AVM at least 30% of CT Angiography (CTA) criteria during the first year of the study (comparison of the volume of the AVM a year versus pre-inclusion).

SECONDARY OUTCOMES:
Treatment efficacy at M3 | After 3 months of treatment
Treatment efficacy at M6 | After 6 months of treatment
Treatment efficacy at M9 | After 9 months of treatment
Treatment tolerability | One year
  Number and description of serious advent events
Treatment Impact on Quality of life | Before treatment initiation and after 12 months of treatment
  Quality of life will be assessed before and at the end of the first year of treatment using a questionnaire given to patients. There is no questionnaire specifically tailored to vascular malformations in the literature. Thus the investigators adapted a document based on an evaluation of the quality of life for survivors of burn injury.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DEVAUCHELLE, MD, PhD, Study Director — CHU Amiens; Emmanuel MORELON, MD, PhD, Study Chair — HCL Lyon
Locations (13):
- UCL, Brussels, Belgium
- France (12):
  - CHU Amiens, Amiens
  - CHU Bordeaux, Bordeaux
  - CHU Dijon, Dijon
  - CHRU Lille, Lille
  - HCL Lyon, Lyon
  - APHM, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nice, Nice
  - APHP, Paris
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No